CLINICAL TRIAL: NCT05336864
Title: Association of Intraoperative Blood Pressure Excursions Below Cerebral Autoregulatory Boundaries With Organ Injury Following Major Noncardiac Surgery (AUTOREGULATE-NONCARDIAC)
Brief Title: Association of Intraoperative Blood Pressure Excursions Below Cerebral Autoregulatory Boundaries With Organ Injury Following Major Noncardiac Surgery
Acronym: AR-NONCARDIAC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-00298; am22Wanner
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Intraoperative Arterial Hypotension
Keywords: cerebral autoregulation; major cardiovascular, renal and neurological complications; hypotension; perioperative myocardial injury; perioperative acute kidney injury; neurological injury; Neurofilament Light Chain (NFL); C-reactive protein (CRP); near-infrared spectroscopy (NIRS)
MeSH Terms: conditions — Hypotension; Trauma, Nervous System; Charcot-Marie-Tooth disease, Type 1F

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-invasive cerebral oximetry monitoring — Main study (all patients): Continuous bilateral frontal cerebral near-infrared spectroscopy (NIRS) monitoring will be performed in all patients for the duration of general anesthesia. Intraoperative parameters including NIRS and invasive blood pressure will be collected and recorded in real-time using the software ICM+.
  Postoperative hemodynamics substudy (facultative): Cerebral NIRS monitoring will be continued postoperatively in a subset of patients being admitted to the ICU.
Other: additional perioperative blood sampling — Main study (all patients): Creatinine, high-sensitivity troponin (T hs-cTnT), Growth/Differentiation Factor-15 (GDF-15), Hemoglobin
  Neurological injury substudy (facultative): Neurofilament Light Chain (NFL) and C-reactive protein (CRP)
Other: clinical & telephone assessments — Main study (all patients): Telephone follow-up (1-year outcomes).
Other: Non-invasive somatic oximetry monitoring — Tissue perfusion substudy (facultative): Continuous somatic NIRS monitoring of an extremity (i.e. on skin of leg or arm) will be performed intraoperatively and postoperatively in a subset of patients being admitted postoperatively to the ICU.
Other: Processed electroencephalogram (pEEG) monitoring — Processed EEG substudy to explore the relationship between processed EEG-derived depth of anesthesia metrics and cerebral autoregulatory function.

SUMMARY:
The aim of study is to investigate the clinical relevance of blood pressure (BP) excursions below cerebral autoregulatory boundaries in major noncardiac surgery. The study seeks to establish a precedent for a personalized definition of intraoperative arterial hypotension based on non-invasive tissue oxygenation measurements. The feasibility of NIRS-based autoregulation monitoring in major noncardiac surgery and the prognostic relevance of BP excursions below the NIRS-derived lower limit of autoregulation (LLA) with regard to major cardiovascular, renal and neurological complications will be investigated.

DETAILED DESCRIPTION:
Major adverse cardiovascular events (MACE) are leading causes of perioperative morbidity and mortality following major noncardiac surgery. Intraoperative arterial hypotension is strongly associated with postoperative morbidity and mortality. However, interventional trials have been unable to demonstrate clinically relevant reductions in the incidence of postoperative MACE, which can potentially be explained by the hitherto lacking consideration of patient-specific autoregulatory boundaries. This is especially problematic considering that the presumed mechanism of hypotension-induced organ injury is hypoperfusion due to transgression of the lower limit of blood flow autoregulation. In other clinical settings, excursions below the autoregulatory threshold have been shown to be superior predictors of adverse events than excursions below absolute blood pressure (BP) thresholds, however, there is a paucity of data in major noncardiac surgery.

This prospective, multicenter cohort observation study aims to investigate the clinical relevance of blood pressure excursions below autoregulatory boundaries and to determine the association of other measures of disturbed intraoperative cerebral autoregulatory function in major noncardiac surgery.

This project will consist of a Main study in which all patients will be enrolled and of substudies on perioperative neurologic injury, tissue perfusion, postoperative hemodynamics, and processed electroencephalogram (EEG), in which selected patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria (All patients):

* undergoing major noncardiac surgery in general anesthesia will be included. Major noncardiac surgery is defined as:

  * vascular surgery (with the exception of arteriovenous shunt, vein stripping procedures and carotid endarterectomies)
  * intraperitoneal surgery
  * intrathoracic surgery
  * major orthopedic surgery
* at cardiovascular risk, defined as meeting at least 1 of the following 6 criteria:

  * preoperative NT-proBNP ≥ 200 ng/l
  * history of coronary artery disease
  * history of peripheral vascular disease
  * history of stroke
  * undergoing major vascular surgery, with the exception of arteriovenous shunt, vein stripping procedures and carotid endarterectomies
  * fulfillment of any 3 of the 8 following criteria:

    * undergoing major surgery (intrathoracic, intraperitoneal or suprainguinal vascular surgery)
    * any history of CHF or history of pulmonary edema
    * anamnestic transient ischemic attack (TIA)
    * diabetes under treatment with either oral antidiabetic agent or insulin
    * age > 70 years
    * history of hypertension
    * serum creatinine > 175 mcmol/l or calculated creatinine clearance < 60 l/min/1.73m2 (Cockroft Gault)
    * history of smoking within 2 years of surgery
* intraoperative continuous invasive blood pressure monitoring indicated due to anesthetic or surgical factors
* planned surgical time ≥ 90 minutes
* planned postoperative hospital stay at least 1 night

Additional inclusion criteria for neurologic injury sub-study:

* Age ≥ 65 years

Exclusion Criteria (All patients):

* pregnancy (anamnestic)
* emergent surgery
* urological surgery
* renal insufficiency with creatinine clearance < 30 ml/min (Cockroft- Gault equation) or on dialysis
* inclusion in an interventional clinical trial with any common endpoints: acute kidney injury, perioperative myocardial injury, components of the composite major cardiovascular, renal and neurological complications up to 1 year following surgery (ACS, CHF, coronary revascularization, stroke, new CKD or progression of CKD, new need for renal replacement therapy, mortality), neurological injury, delirium, exception: potential inclusion of subset of patients in RCT investigating the perioperative use of colchicine in major noncardiac surgery (COLCAT study).
* previously enrolled in this study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be screened for eligibility during the preoperative anesthetic visit based on the inclusion/exclusion criteria and the previous medical history using a standardized checklist, helping to minimize bias.
Sampling Method: Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Perioperative organ injury on postoperative days 1-3, a composite of: | postoperative days 1-3
  o perioperative myocardial injury (defined as an absolute perioperative rise in high-sensitivity troponin T [hsTnT] of ≥ 14 ng/l above preoperative values or between two postoperative measurements, if preoperative hs-cTnT is missing)
  and/or
  o perioperative acute kidney injury (defined as absolute perioperative increase in serum creatinine of > 26.4 μmol/l or a percentage perioperative increase in serum creatinine of > 50%)

SECONDARY OUTCOMES:
Major cardiovascular, renal and neurological complications up to 1 year following surgery, a composite of any of the following: | up to 1 year following surgery
  * acute coronary syndrome
  * acute congestive heart failure (CHF)
  * coronary revascularization
  * stroke
  * new or progressive chronic kidney disease (CKD)
  * new need for renal replacement therapy (RRT)
  * all-cause mortality
  * cardiovascular mortality
Neurological injury (neurological injury sub-study) | postoperative day 2
  Perioperative trajectory of serum neurofilament light chain (NFL)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M Wanner, Dr. med., Principal Investigator — Clinic for Anaesthesia, University Hospital Basel
Locations (3):
- Switzerland (3):
  - University Hospital Basel, Clinic for Anaesthesia, Intermediate Care, Prehospital Emergency Medicine and Pain Therapy, Basel
  - Inselspital, Bern University Hospital, Department of Anaesthesiology and Pain Medicine, Bern
  - Cantonal Hospital St. Gallen, Division of Perioperative Intensive Care Medicine, Sankt Gallen